CLINICAL TRIAL: NCT01129466
Title: Effects of Sulforaphane Containing Supplements on Nasal Cell Phase 2 Gene Expression in Healthy Volunteers.
Brief Title: Effects of 2 Different Broccoli Sprout Containing Supplements on Nasal Cells in Healthy Volunteers
Acronym: Broccosprout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Terry Noah, MD, Principal Investigator, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 10-0410; 1R01HL095163-01A2 (NIH)
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Healthy Adult Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplement A followed by supplement B (Active Comparator)
  Interventions: Dietary Supplement: Supplement A followed by Supplement B
- Supplement B followed by Supplement A (Active Comparator)
  Interventions: Dietary Supplement: Supplement B followed by Supplement A

INTERVENTIONS:
Dietary Supplement: Supplement A followed by Supplement B — Supplement A (3 days of Broccosprout homogenate) will be followed at least 2 weeks later by Supplement B (3 days of Broccosprout sandwich and SFN rich tea)
  Arms: Supplement A followed by supplement B
Dietary Supplement: Supplement B followed by Supplement A — Supplement B (Broccosprout sandwich and SFN rich tea for 3 days) followed at least 2 weeks later by 3 days of Supplement A (Broccosprout homogenate)
  Arms: Supplement B followed by Supplement A

SUMMARY:
Purpose: To compare the change in nasal cell HO-1 expression induced by two different preparations of sulforaphane (SFN)-containing nutritional supplements Participants: Healthy nonsmoking young adults, age 18-35 Procedures (methods): This pilot study will use a randomized crossover design. Subjects will be randomized to receive either the equivalent of 4 ounces/day of fresh broccoli sprouts (FBS) in food and tea, or the equivalent amount as broccoli sprout homogenates (BSH), for 3 consecutive days. Nasal lavage and blood samples will be obtained before, during and after this 3-day period. After at least a 2-week washout interval, the protocol will be repeated with the alternate supplement. The primary analysis will test the hypothesis that broccoli sprouts in food will increase HO-1 expression to a similar degree as the equivalent amount of sprouts in BSH

DETAILED DESCRIPTION:
Broccoli sprouts are a concentrated source of the potent phase 2 enzyme (antioxidant) potentiator, sulforaphane (SFN) in the form of its natural precursor, sulforaphane glucosinolate (SGS™). SFN is an isothiocyanate which has generated interest recently as a chemopreventive agent in cancer research, and as an antioxidant in inflammation research. Recently published data show that 3 days intake of broccoli sprouts in homogenate form is followed by significant upregulation of several phase 2 enzymes in nasal cells. Our group's research at the UNC Center for Environmental Medicine, Asthma and Lung Biology (CEMALB) focuses on the effects of oxidant pollutants on inflammatory and host defense responses to viral infections. One of the aims of our grant is to measure the effects of pre-treatment with SFN supplements, on nasal responses to live attenuated influenza virus vaccines. In preparation for this larger study, we here propose a pilot study comparing the effects of the published BSH supplement, vs. supplementation with foods containing fresh broccoli sprouts, on relevant nasal endpoints and serum SFN levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, nonsmoking adults, age 18-35 yr
* Willing to avoid cruciferous vegetables for 1 week prior to study entry and for 2 sets of the 4 study sessions

Exclusion Criteria:

* Inability/unwillingness to avoid anti-inflammatory medications (inhaled, topical or systemic) prior to and during the study. Duration of prohibition prior to study will based on drug half life x 6 (ie 1 day for ibuprofen, 4 days for naproxen etc);
* Inability/unwillingness to avoid antioxidant vitamins and juices or drinks with vitamin supplements added for 2 days prior to enrollment and throughout the study;
* History or symptoms of allergic rhinitis;
* Respiratory infection (cough, sore throat, sinusitis, fever etc) within prior 4 weeks;
* Current nutritional disorder such as anorexia, bulimia, irritable bowel syndrome, Crohn's disease etc;
* Pregnancy or nursing;
* Asthma (other than wheezing occurring only in childhood); immunodeficiency (HIV or other); or any chronic medical condition that, in the opinion of the investigator, would preclude subject participation;
* Current use of immunosuppressive drugs including corticosteroids.
* Lactose and/or gluten deficiency
* History of fainting or feeling severely dizzy with blood draws

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
the change in nasal cell HO-1 expression induced by two different preparations of sulforaphane (SFN)-containing nutritional supplements | 2 hours

SECONDARY OUTCOMES:
serum SFN level | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Terry Noah, MD, Principal Investigator — University of North Carolina at Chapel Hill, Dept of Pediatrics / Center for Environmental Medicine, Asthma and Lung Biology
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States